CLINICAL TRIAL: NCT02397941
Title: Diastasis Recti Abdominis and Abdominal Muscles in Pregnant and Non-pregnant Women
Brief Title: Diastasis Recti Abdominis and Abdominal Muscles
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr.2015-0008
Record Dates: First submitted 2015-03-13; First posted 2015-03-25 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Interrectal Distance; Diastasis Recti; Dimensions of the Muscles of the Lateral Abdominal Wall
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- non-pregnant women: 20 non-pregnant women, BMI < 30 kg/m2, Nulligravidas, no abdominal pre-operations, aged 20-45 years, measurement of the abdominal muscles and interrectal distance by ultrasound
  Interventions: Other: Ultrasound
- pregnant women: 40 pregnant women, BMI < 30 kg/m2 before pregnancy, Primigravidas, no abdominal pre-operations, aged 20-45 years, measurement of the abdominal muscles and interrectal distance by ultrasound, consecutive measurement during the course of pregnancy
  Interventions: Other: Ultrasound
- women who deliverd: 20 pregnant women, BMI < 30 kg/m2 before pregnancy, Primiparas, no abdominal pre-operations, aged 20-45 years, measurement of the abdominal muscles and interrectal distance by ultrasound, measurement after delivery (10 after spontaneous delivery, 10 after elective cesarean section)
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — ultrasound measures

SUMMARY:
Purpose of the study is the assessment of interrectal distance and dimensions of the muscles of the lateral abdominal wall in pregnant and non-pregnant women

DETAILED DESCRIPTION:
* Purpose of the study is the assessment of interrectal distance and dimensions of the muscles of the lateral abdominal wall in pregnant and non-pregnant women
* Assessment via ultrasound measurement transabdominally
* 3 groups of participants: 1.) 20 pregnant women, who have never been pregnant before; 2.) 40 pregnant women with their first pregnancy, followed over the course of pregnancy; 3.) 20 women1-5 days after delivery (10 after spontaneous delivery, 10 after planned cesarean section)
* comparison between pregnant and non-pregnant women; evaluation of influence of pregnancy and mode of delivery

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant women aged 20-45 y with a BMI < 30 kg/m2 who never were pregnant
* pregnant women aged 20-45 y with a BMI < 30 kg/m2 before pregnancy

Exclusion Criteria:

* abdominal pre-operations
* chronical lung diseases
* constipation
* maternal collagenosis
* polyhydramnion (AFI > 25)
* uterus fibroids > 10 cm
* inability to perform Valsalva

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion:
  * non-pregnant women aged 20-45 y with a BMI < 30 kg/m2 who never were pregnant
  * pregnant women aged 20-45 y with a BMI < 30 kg/m2 before pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
interrectal distance | baseline

SECONDARY OUTCOMES:
measurement of the abdominal muscles of the lateral abdominal wall by ultrasound. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nina Kimmich, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland